CLINICAL TRIAL: NCT03876990
Title: Clinical and Medico-economic Evaluation of a Rapid Test (ePlex-BCID®, GenMark) for the Diagnosis of Bacteremia or Fungemia From Positive Blood Culture Bottles, Combining Fast Identification of Bacteria and Fungi and Evaluation of Bacterial Resistance to First Line Antibiotics.
Brief Title: Clinical and Medico-economic Evaluation of a Rapid Test (ePlex-BCID®, GenMark) for the Diagnosis of Bacteremia and Fungemia.
Acronym: HEMOFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: GenMark Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 38RC15.091
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Bacteremia Sepsis; Fungemia
Keywords: multiplex PCR; blood culture; rapid diagnosis
MeSH Terms: conditions — Fungemia

STUDY DESIGN:
Intervention Model Description: Randomized assignation. Half of the patients will be diagnosed by the rapid test in addition to current diagnosis strategy and the other half by current diagnosis strategy alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multiplex PCR + Current strategy (Experimental): Results of the multiplex PCR will be send as soon as possible to the infectious disease phycian for quick adaptation of antibiotic treatment. Positive blood cultures will also undergo current diagnosis strategy for bacteremia and fungemia.
  Interventions: Diagnostic Test: Multiplex PCR
- Current strategy alone (Active Comparator): Current diagnostic strategy based on the identification of bacteria and micromyces isolated in blood cultures after subculture by mass spectrometry (MALDI-TOF) and determination of their sensitivity to antibiotics or antifungals by antibiotic susceptibility testing or antifungigram
  Interventions: Diagnostic Test: Current strategy alone

INTERVENTIONS:
Diagnostic Test: Multiplex PCR — Quick adaptation of antibiotic treatment according to the species identified and to the results of the resistance markers present in the multiplex PCR
  Arms: Multiplex PCR + Current strategy
Diagnostic Test: Current strategy alone — Identification of bacteria and micromyces isolated in blood cultures after subculture by mass spectrometry (MALDI-TOF) and determination of their sensitivity to antibiotics or antifungals by antibiotic susceptibility testing or antifungigram
  Other Names: MALDI-TOFF identification
  Arms: Current strategy alone

SUMMARY:
This study evaluates the clinical benefit of a rapid test for fast diagnosis of bacteremia and fungemia from positive blood cultures in case of sepsis. This assay enables rapid identification of bacteria and fungi and allows to evaluate bacterial resistance to first line antibiotics. The clinical and medico-economic impact of this assay used in addition to the current diagnosis strategy (half of the patients) will be compared to the current diagnostic strategy alone (other half of the patient).

DETAILED DESCRIPTION:
Bacteremia and fungemia are severe complications, sometimes life-threatening, of every sepsis. During septicemia, every hour matters to start an appropriate antibiotic or antifungal treatment as every hour of delay is associated to higher death rate.

The rapid multiplex PCR assay that is evaluated in this study allows to identify in 60 to 90 minutes, the bacteria or fungi that is present in the positive blood culture bottles and to identify resistance markers to first line antibiotics that are used to treat sepsis. This strategy allows quicker adaptation of antibacterial or antifungal treatment based on the species of the bacteria or fungi identified and on the results of the resistance markers compared to current diagnosis strategy of bacteremia or fungemia. This quicker adaptation could lead to improved survival rate, reduced complications of sepsis, reduced hospital stay length and could reduce the use of large spectrum antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bacteremia and/or fungemia defined by :

  1/ the presence of clinical signs of sepsis; AND 2/ a positive blood culture, i.e. the growth of at least one species of bacteria or micromyces in at least one blood culture vial
* Patient Hospitalized at Grenoble University Hospital (only North site) and seen by a physician from the antibiotic stewardship team
* First blood culture positive for the patient's sepsis episode
* Informed and written consent signed by the patient or his legal representative or the doctor in case of emergency.

Exclusion Criteria:

* Patients mentioned in the law articles L1121-5 to L1121-8 from French Health Code
* Patients hospitalized in palliative care unit
* Persons with an estimated survival of less than one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Delay from suspicion of sepsis to optimized antibiotic/antifungal treatment | Follow up is set to hospital length stay with a maximum of 30 days
  Delay between first sampling of blood cultures for sepsis and optimized antibiotic/antifungal treatment. Treatment will be considered optimized if it is active on the bacteria/fungi responsible for sepsis and if it follows current treatment recommendations for the bacteria/fungi identified.

SECONDARY OUTCOMES:
Medical evaluation of the consequences of the innovative strategy compared to current strategy : 30-day mortality | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : 30-day mortality
Medical evaluation of the consequences of the innovative strategy compared to current strategy : complication rate | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : complication rate (ICU admission or length of stay, antibiotic/antifungal treatment toxicity rate, recurrence of sepsis within 30 days, re-admission to hospital within 30 days)
Medical evaluation of the consequences of the innovative strategy compared to current strategy : length of hospital stay | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : length of hospital stay
Medical evaluation of the consequences of the innovative strategy compared to current strategy : antibiotic treatment duration | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : treatment duration for antibiotics with high impact on the commensal flora (i.e. : carbapenems) or with high toxicity (i.e. : vancomycin)
Medical evaluation of the consequences of the innovative strategy compared to current strategy : delay of antibiotic/antifungal treatment modification at several time points | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : delay of antibiotic/antifungal treatment modification at several time points (after the result of the Gram stain, after the results of the multiplex PCR, after the results of the identification of the bacteria/fungi and after the results of antibiotic/antifungal treatment susceptibility).
Medical evaluation of the consequences of the innovative strategy compared to current strategy : rate of antibiotic/antifungal treatment modification at several time points | Hospital length stay with a maximum of 30 days
  The following clinical consequences will be measured and compared in each arm : rate of antibiotic/antifungal treatment modification at several time points (after the result of the Gram stain, after the results of the multiplex PCR, after the results of the identification of the bacteria/fungi and after the results of antibiotic/antifungal treatment susceptibility).
Economic evaluation of the hospitalization costs of the innovative strategy compared to current strategy | Hospital length stay with a maximum of 30 days
  Hospitalization costs will be measured
Economic evaluation of the treatments costs of the innovative strategy compared to current strategy | Hospital length stay with a maximum of 30 days
  Anti-infectious treatment costs will be measured
Economic evaluation of the costs of the innovative compared to current strategy | Hospital length stay with a maximum of 30 days
  Costs of the innovative assay (reagents and device) will be measured
Economic evaluation of the medical imaging costs of the innovative strategy compared to current strategy | Hospital length stay with a maximum of 30 days
  Medical imaging costs will be measured
Economic impact of the introduction of the innovative strategy for Grenoble University Hospital | Extrapolation of the costs for a one year period
  Measurement and evaluation of the economic impact of the innovative strategy on the budget of Grenoble University Hospital, on the target population, for a period of one year.

CONTACTS AND LOCATIONS:
Overall Officials: Yvan CASPAR, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Huang TD, Melnik E, Bogaerts P, Evrard S, Glupczynski Y. Evaluation of the ePlex Blood Culture Identification Panels for Detection of Pathogens in Bloodstream Infections. J Clin Microbiol. 2019 Jan 30;57(2):e01597-18. doi: 10.1128/JCM.01597-18. Print 2019 Feb. PMID 30487304
- [Background] Banerjee R, Teng CB, Cunningham SA, Ihde SM, Steckelberg JM, Moriarty JP, Shah ND, Mandrekar JN, Patel R. Randomized Trial of Rapid Multiplex Polymerase Chain Reaction-Based Blood Culture Identification and Susceptibility Testing. Clin Infect Dis. 2015 Oct 1;61(7):1071-80. doi: 10.1093/cid/civ447. Epub 2015 Jul 20. PMID 26197846
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Patel TS, Kaakeh R, Nagel JL, Newton DW, Stevenson JG. Cost Analysis of Implementing Matrix-Assisted Laser Desorption Ionization-Time of Flight Mass Spectrometry Plus Real-Time Antimicrobial Stewardship Intervention for Bloodstream Infections. J Clin Microbiol. 2016 Dec 28;55(1):60-67. doi: 10.1128/JCM.01452-16. Print 2017 Jan. PMID 27795335
- [Background] Maubon D, Dard C, Garnaud C, Cornet M. Profile of GenMark's ePlex(R) blood culture identification fungal pathogen panel. Expert Rev Mol Diagn. 2018 Feb;18(2):119-132. doi: 10.1080/14737159.2018.1420476. Epub 2017 Dec 28. PMID 29284316
- [Background] Timbrook TT, Morton JB, McConeghy KW, Caffrey AR, Mylonakis E, LaPlante KL. The Effect of Molecular Rapid Diagnostic Testing on Clinical Outcomes in Bloodstream Infections: A Systematic Review and Meta-analysis. Clin Infect Dis. 2017 Jan 1;64(1):15-23. doi: 10.1093/cid/ciw649. Epub 2016 Sep 26. PMID 27678085